CLINICAL TRIAL: NCT00058812
Title: Administration of EBV Specific Cytotoxic T Lymphocytes to Recipients of Mismatched-Related or Phenotypically Similar Unrelated Donor Marrow Grafts
Brief Title: Giving Epstein-Barr Virus (EBV) Specific Killer T Lymphocytes to Patients Who Have Had Donor Marrow Grafts
Acronym: ETNA
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: The Methodist Hospital Research Institute (Other); Center for Cell and Gene Therapy, Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Helen Heslop, Professor, Baylor College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 6676-ETNA; ETNA; NCT00608309 (obsolete NCT alias)
Record Dates: First submitted 2003-04-11; First posted 2003-04-15 (Estimated); Last update posted 2015-01-29 (Estimated); Status verified 2015-01

CONDITIONS: Epstein-Barr Virus Infections
Keywords: Cytotoxic T Lymphocytes; bone marrow transplant; EBV+ lymphoproliferative disease
MeSH Terms: conditions — Epstein-Barr Virus Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- EBV specific T cells (Experimental): EBV specific T cells
  Interventions: Biological: EBV specific T cells

INTERVENTIONS:
Biological: EBV specific T cells — One injection of 2x10^7 cells/m2 from Day 45 post transplant. If EBV DNA levels remain elevated above 1000 copies/ug or the patient has persistent disease they will be eligible to receive up to 5 additional injections of CTLs at the original dose at monthly intervals.

SUMMARY:
Patients have a type of blood cell cancer or other blood problem that is very hard to cure with standard treatments and s/he will receive a bone marrow transplant. If the patient does not have a brother or sister whose marrow is a "perfect match", this bone marrow will come from a donor whose marrow is the best match available. This person may be a close relative or an unrelated person whose bone marrow best "matches" the patient's, and who agrees to donate marrow.

In normal people, the Epstein-Barr (EB) virus infection causes a flu like illness and usually gets better when the immune system controls the infection. The virus, however, remains hidden in the body for life. After a transplant, while the new immune system is growing back, the EB virus can come out and infect cells and cause them to grow in an uncontrolled manner. Patients can develop fevers, swollen lymph nodes and damage to other organs such as kidneys and lungs. This infection acts like a cancer because the cells infected with EB virus grow very quickly and there is no known effective treatment. This sort of infection will occur in between 10-30% of patients receiving a transplant from a donor who is not a perfect match, and has been fatal in nearly all these cases.

This infection occurs because the immune system cannot control the growth of the cells. We want to see if we can prevent it from happening or treat it by giving the patient a kind of white blood cell called T cells that we have grown from the marrow donor. These cells have been trained to attack EB virus infected cells. We will grow these T cells from blood taken from the donor at the time of bone marrow harvest. These T cells will be stimulated with the donor's EB virus-infected cells which have been treated with radiation so they cannot grow. After mixing these cells together we will be able to grow special T cells from the donor that can attack EB virus infected cells. We will then collect the T cells and make sure they can kill the virus infected cells. These EBV specific T cells are an investigational product not approved by the Food and Drug Administration.

DETAILED DESCRIPTION:
We will obtain blood from the donor and will first make a B cell line called a lymphoblastoid cell line or LCL by infecting the blood with a laboratory strain of EBV called B95. We will then use this EBV-infected cell line (which have been treated with radiation so that they cannot grow) as stimulator cells and mix it with more blood. This stimulation will train the T cells to kill EBV infected cells and result in the growth of an EBV specific T cell line. We will then test the T cells to make sure that they kill the EBV infected cells and not the normal cells and freeze them.

The marrow donor's T cells will be thawed and injected through an intravenous line for a period of 10 minutes. The subject may be premedicated with diphenhydramine (Benadryl) and acetaminophen (Tylenol). We would give one dose of the cells on or after day 45 following transplant if the subject agreed and was well enough. If the EBV DNA levels remain high or the subject has persistent disease, s/he may be eligible to receive up to 5 additional injections of T cells at the original dose at monthly intervals. After the subject has received the T cells, s/he will be contacted by the research nurse or another member of the study team weekly for 6 weeks, then once every three months for a year so that we can check on his/her progress.

We will continue to follow the subject in the BMT clinic after the injections. To learn more about the way the T cells are working, an extra 40 mls (about 8 teaspoonfuls) of blood will be taken pre-infusion, 4 hours after the infusion, 3-4 days post infusion (optional) and at 1, 2, 4 and 6 weeks after the T cell infusions, and then at 3, 6, 9, and 12 months post infusion. The blood should come from the central intravenous line, and should not require extra needle sticks.

ELIGIBILITY:
INCLUSION CRITERIA:

* All patients receiving a T cell depleted BMT from a mismatched family member or unrelated donor will be eligible for this protocol. In addition, patients receiving a matched sibling transplant or T replete transplant may be eligible if they are at high risk of developing EBV LPD because of their underlying disease (e.g Wiskott-Aldrich or Ataxia Telangiectasia) or have a past history of EBVLPD or other EBV associated malignancy.
* O2 saturation > 90% on room air

EXCLUSION CRITERIA:

- Exclusion criteria for BMT will be as detailed in the relevant protocol.

Exclusion criteria at time of administration CTLs:

* Patients with GVHD of Grade II or greater.
* Patients with severe renal disease (i.e., creatinine clearance less than half normal for age).
* Patients with severe hepatic disease (bilirubin greater than twice normal, or SGOT greater than 3 x normal).
* Patients with a severe intercurrent infection.
* Patients with a life expectancy <6 weeks

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 1993-05; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Safety of one intravenous injection of BMT donor derived EBV specific cytotoxic T lymphocytes (CTLs) in BMT recipients at high risk. | 1 year
To compare the antiviral and immunological efficacy of a single dose of CTLs compared to the multiple dose regimens previously employed | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Helen E Heslop, MD, Principal Investigator — Center for Cell and Gene Therapy, Baylor College of Medicine
Locations (2):
- United States (2):
  - Houston Methodist Hospital, Houston, Texas
  - Texas Children's Hospital, Houston, Texas

REFERENCES:
- [Derived] Cohen JI, Jaffe ES, Dale JK, Pittaluga S, Heslop HE, Rooney CM, Gottschalk S, Bollard CM, Rao VK, Marques A, Burbelo PD, Turk SP, Fulton R, Wayne AS, Little RF, Cairo MS, El-Mallawany NK, Fowler D, Sportes C, Bishop MR, Wilson W, Straus SE. Characterization and treatment of chronic active Epstein-Barr virus disease: a 28-year experience in the United States. Blood. 2011 Jun 2;117(22):5835-49. doi: 10.1182/blood-2010-11-316745. Epub 2011 Mar 31. PMID 21454450
- [Derived] Heslop HE, Slobod KS, Pule MA, Hale GA, Rousseau A, Smith CA, Bollard CM, Liu H, Wu MF, Rochester RJ, Amrolia PJ, Hurwitz JL, Brenner MK, Rooney CM. Long-term outcome of EBV-specific T-cell infusions to prevent or treat EBV-related lymphoproliferative disease in transplant recipients. Blood. 2010 Feb 4;115(5):925-35. doi: 10.1182/blood-2009-08-239186. Epub 2009 Oct 30. PMID 19880495